CLINICAL TRIAL: NCT02338518
Title: Comparison of SEEOX and SOX Chemotherapeutic Regimens in Stage ⅢB/ⅢC Gastric Cancer Patients
Brief Title: Comparison of SEEOX and SOX Regimens in Stage ⅢB/ⅢC Gastric Cancer Patients
Acronym: SVOSA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Li Guoli, professor, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20140621; 08Z28 (Other Grant/Funding Number: Nanjing Military Region)
Record Dates: First submitted 2014-10-15; First posted 2015-01-14 (Estimated); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Stomach Neoplasms; Gastric Cancer
Keywords: gastric cancer; neoadjuvant chemotherapy; efficacy; safety
MeSH Terms: conditions — Stomach Neoplasms | interventions — Oxaliplatin; Etoposide; Epirubicin; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SEEOX group (Experimental): A three-cycle neo-adjuvant chemotherapy was performed in all cases. In every cycle, oxaliplatin 100 mg/m2, etoposide 80 mg/m2, and pharmorubicin 30 mg/m2 were administered from the celiac artery on day 1. 80～120 mg of oral S-1 per square meter of body-surface area per day was given for 2 weeks. The second cycle was scheduled following a 1-week rest after the first cycle.
  Interventions: Drug: oxaliplatin; Drug: etoposide; Drug: pharmorubicin; Drug: S-1
- SOX group (Active Comparator): A three-cycle neo-adjuvant chemotherapy was performed in all cases. In every cycle, patients received intravenous oxaliplatin 130 mg/m2 on day 1, and 80~120 mg of oral S-1 per square meter of body-surface area per day was given for 2 weeks. The second cycle was scheduled following a 1-week rest after the first cycle.
  Interventions: Drug: oxaliplatin; Drug: S-1

INTERVENTIONS:
Drug: oxaliplatin — oxaliplatin 100 mg/m2 was administered from the celiac artery on day 1 of every cycle in SEEOX group and SOX group.
  Intravenous oxaliplatin 130 mg/m2 was administered on day 1 of every cycle in SOX group.
Drug: etoposide — etoposide 80 mg/m2 was administered from the celiac artery on day 1 of every cycle in SEEOX group.
  Arms: SEEOX group
Drug: pharmorubicin — pharmorubicin 30 mg/m2 was administered from the celiac artery on day 1 of every cycle in SEEOX group.
  Other Names: epirubicin
  Arms: SEEOX group
Drug: S-1 — 80~120 mg of oral S-1 per square meter of body-surface area per day was given for 2 weeks in both SEEOX and SOX groups.

SUMMARY:
Chemotherapy is an important therapeutic method for patients with advanced gastric cancer. However, there is currently no established standard chemotherapeutic regimen in the preoperative or neoadjuvant treatment setting. The aim of our study was to compare the efficacy and toxicity between SEEOX and SOX regimens. The investigators estimate that combined intravenous and intra-arterial intensified SEEOX preoperative chemotherapy may be a safe and promising regimen for locally advanced or initially unresectable gastric cancer patients.

DETAILED DESCRIPTION:
Gastric cancer patients who will receive neoadjuvant chemotherapy would be included in this study. They would receive combined intravenous and intra-arterial intensified SEEOX neoadjuvant chemotherapy or SOX regimen at random. The efficacy and toxicity of these two regimens would be compared.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group(ECOG) score 0-2
* Ambulatory males or females, aged 30-70 years.
* Unresectable gastric cancer (Tumors with bulky nodal metastases surrounding the celiac artery and its branches or invasion of adjacent structures such as pancreas, omentum, esophagus, and aorta were considered unresectable)
* Life expectancy more than 3 months
* Give written informed consent, with the understanding that the patient has the right to withdraw from the study at any time, without prejudice.
* Normal hepatic, renal, and bone marrow function (GPT<2 fold of upper limit value; white blood cell count>4000/dl, Tbil<1.5mg/dl, Cr<1.5 fold of upper limit value)

Exclusion Criteria:

* Patients can not bear surgical procedure.
* Pregnant or lactating women.
* Previous cytotoxic chemotherapy, radiotherapy or immunotherapy.
* History of another malignancy within the last five years.
* History of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the Investigator to be clinically significant precluding informed consent or interfering with compliance for oral drug intake.
* Clinically significant (i.e. active) cardiac disease e.g. symptomatic coronary artery disease, New York Heart Association (NYHA) grade II or greater congestive heart failure or serious cardiac arrhythmia requiring medication or myocardial infarction within the last 12 months.
* Organ allografts requiring immunosuppressive therapy.
* Serious uncontrolled intercurrent infections or other serious uncontrolled concomitant disease.
* Moderate or severe renal impairment: serum creatinine > 1.5 x upper limit of normal (ULN).
* Hypersensitivity to any drug of the study regimen.
* With abdominal cavity implantation metastasis or distant metastasis.
* Unwilling or unable to comply with the protocol for the duration of the study.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2015-01-04 (Actual); Primary Completion 2019-05-21 (Actual); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
3 year progression free survival | up to 7 years
  time period calculated from randomization to the first disease progression, recurrence or death from any cause

SECONDARY OUTCOMES:
Objective response rate | up to 4 years
  the proportion of patients with complete and partial response according to Response Evaluation Criteria in Solid Tumors guidelines (version 1.1)
R0 resection rate | up to 4 years
  the proportion of complete tumor resection with no microscopic or macroscopic residual diseases in all operations
3 year overall survival | up to 7 years
  time period calculated from randomization to death from any cause
Adverse events of preoperative chemotherapy | up to 4 years
  preoperative chemotherapy associated complications

OTHER OUTCOMES:
Sensitivity analysis of primary outcome adjusted for stratification factors | up to 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Guoli Li, M.D., Study Chair — Jinlin Hospital
Locations (1):
- Jinling Hospital, Nanjing, Jiangsu, China